CLINICAL TRIAL: NCT00904202
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Of Lidocaine Patch 5% Alone, Gabapentin Alone, And Lidocaine Patch 5% And Gabapentin In Combination For The Relief Of Pain In Patients With Diverse Peripheral Neuropathic Pain Conditions
Brief Title: A Study Of Lidocaine Patch 5% Alone, Gabapentin Alone, And Lidocaine Patch 5% And Gabapentin In Combination For The Relief Of Pain In Patients With Diverse Peripheral Neuropathic Pain Conditions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr Director, Clinical R&D, Endo Pharmaceuticals Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3220-009
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Postherpetic Neuralgia; Diabetic Neuropathy; Complex Regional Pain Syndrome; Carpal Tunnel Syndrome; HIV Neuropathy; Idiopathic Sensory Neuropathy; Peripheral Neuropathy
MeSH Terms: conditions — Neuralgia, Postherpetic; Diabetic Neuropathies; Complex Regional Pain Syndromes; Carpal Tunnel Syndrome; Peripheral Nervous System Diseases | interventions — Lidoderm; Gabapentin; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo capsules + placebo patch (Placebo Comparator): Placebo to match lidocaine patch; up to four patches applied topically once daily (q24h) to the area of maximal peripheral pain AND Placebo capsules to match gabapentin for oral dosing
  Interventions: Drug: Placebo Capsules + Placebo Patch
- placebo capsules + Lidoderm patch (Lidocaine Group) (Experimental): Lidoderm (lidocaine patch 5%), up to four patches applied topically once daily (q24h) to the area of maximal peripheral pain AND Placebo capsules to match gabapentin for oral dosing
  Interventions: Drug: Placebo capsules + Lidoderm®
- Gabapentin capsules 1800 mg/day + placebo patch (Active Comparator): Gabapentin 300 mg capsules for oral dosing at a dose of 1800 mg/day AND Placebo patch to match lidocaine patch; up to four patches applied topically daily (q24h) to the area of maximal peripheral pain
  Interventions: Drug: Gabapentin + Placebo; Drug: Gabapentin 300 mg capsules 1800 mg/day + placebo patch
- Gabapentin capsules 1800 mg/day + Lidoderm patch (Other): Gabapentin 1800 mg/day AND Lidoderm (lidocaine patch 5%), up to four patches applied topically once daily (q24h) to the area of maximal peripheral pain
  Interventions: Drug: Gabapentin + Lidoderm®; Drug: Gabapentin 1800 mg/day + Lidoderm patch

INTERVENTIONS:
Drug: Placebo Capsules + Placebo Patch — Patients participated in a 5-week treatment period. Eligible patients were randomized into one of four treatment groups: placebo capsules + placebo patch (Placebo Group), placebo capsules + Lidoderm patch (Lidocaine Group), Gabapentin capsules 1800 mg/day + placebo patch (Gabapentin Group), or Gabapentin capsules 1800 mg/day + Lidoderm patch (Combination Group).
  Other Names: Lidocaine patch 5%
  Arms: placebo capsules + placebo patch
Drug: Placebo capsules + Lidoderm® — Patients participated in a 5-week treatment period. Eligible patients were randomized into one of four treatment groups: placebo capsules + placebo patch (Placebo Group), placebo capsules + Lidoderm patch (Lidocaine Group), Gabapentin capsules 1800 mg/day + placebo patch (Gabapentin Group), or Gabapentin capsules 1800 mg/day + Lidoderm patch (Combination Group).
  Other Names: Lidocaine patch 5%
  Arms: placebo capsules + Lidoderm patch (Lidocaine Group)
Drug: Gabapentin + Placebo — Patients participated in a 5-week treatment period. Eligible patients were randomized into one of four treatment groups: placebo capsules + placebo patch (Placebo Group), placebo capsules + Lidoderm patch (Lidocaine Group), Gabapentin capsules 1800 mg/day + placebo patch (Gabapentin Group), or Gabapentin capsules 1800 mg/day + Lidoderm patch (Combination Group).
  Other Names: Lidocaine patch 5%
  Arms: Gabapentin capsules 1800 mg/day + placebo patch
Drug: Gabapentin + Lidoderm® — Patients participated in a 5-week treatment period. Eligible patients were randomized into one of four treatment groups: placebo capsules + placebo patch (Placebo Group), placebo capsules + Lidoderm patch (Lidocaine Group), Gabapentin capsules 1800 mg/day + placebo patch (Gabapentin Group), or Gabapentin capsules 1800 mg/day + Lidoderm patch (Combination Group).
  Other Names: Lidocaine patch 5%
  Arms: Gabapentin capsules 1800 mg/day + Lidoderm patch
Drug: Gabapentin 300 mg capsules 1800 mg/day + placebo patch — Gabapentin 300 mg capsules 1800 mg/day + placebo patch
  Arms: Gabapentin capsules 1800 mg/day + placebo patch
Drug: Gabapentin 1800 mg/day + Lidoderm patch
  Arms: Gabapentin capsules 1800 mg/day + Lidoderm patch

SUMMARY:
Patients with postherpetic neuralgia (PHN), diabetic neuropathy (DN), complex regional pain syndrome (CRPS), carpal tunnel syndrome, HIV neuropathy, idiopathic sensory neuropathy, or other peripheral neuropathy participated in a Phase IV clinical trial to assess the comparative efficacy and safety of Lidoderm monotherapy versus gabapentin monotherapy in treating a diverse group of peripheral neuropathic pain patients.

ELIGIBILITY:
Inclusion Criteria:

1. Had a diagnosis of PHN, DN, CRPS, carpal tunnel syndrome, HIV neuropathy, idiopathic sensory neuropathy, or other peripheral neuropathy (upon mutual agreement of the sponsor and investigator)
2. Patients with PHN must have had pain >3 months after rash healing
3. Patients with DN must have had Type I or II diabetes and painful distal symmetric sensorimotor polyneuropathy with or without dynamic allodynia of the lower extremities
4. Patients with CRPS must have met current IASP (International Association for the Study of Pain) diagnostic criteria
5. Patients with carpal tunnel syndrome must have had a diagnosis by combination clinical neurological examination (e.g., Phalen's and Tinel's signs), electrodiagnostic testing, and daily painful symptoms of at least 3 months' duration
6. Patients with HIV neuropathy must have had HIV, subjective symptoms of painful peripheral neuropathy, and daily painful symptoms of at least 3 months' duration
7. Patients with idiopathic sensory neuropathy must have had pain of at least 3 months' duration
8. Reached an average daily pain rating during the baseline week of pain ratings greater than 4 on the 0-to-10 numerical pain rating scale (Question 5 of the BPI)
9. Had never received an analgesic regimen that contained lidocaine or gabapentin

Exclusion Criteria:

1. Had a neurological condition other than that associated with their pain diagnosis which, in the opinion of the investigator, would interfere with their ability to participate in the study
2. Were taking a lidocaine-containing product that could not be discontinued while receiving lidocaine
3. Were taking class 1 anti-arrhythmic drugs (e.g., mexiletine, tocainide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-01; Primary Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Average daily pain intensity (BPI Questions 3,4,5, and 6) | Visit - V2 (Day 0), V3 (Day 7), V4 (Day 14), V5 (Day 21), V6 (Day 28), V7/EOS (Day 35)

SECONDARY OUTCOMES:
Pain Quality Assessment Scale (PQAS)
Investigator and Patient Global Impression of Change
Allodynia Testing
QoL; Symptom Checklist, pain interference with QoL
Patient Global Impression of Treatment Satisfaction, disability assessment, and Percent Pain Relief (BPI Question 8)
Safety assessments include adverse events; dermal assessments/sensory testing, clinical laboratory tests, vital sign measurements and physical/neurological examination

CONTACTS AND LOCATIONS:
Overall Officials: Sr Director, Study Director — Endo Pharmaceuticals
Locations (7):
- United States (7):
  - Birmingham, Alabama
  - Hueytown, Alabama
  - Phoenix, Arizona
  - Pembroke Pines, Florida
  - New York, New York
  - Rochester, New York
  - Altoona, Pennsylvania